CLINICAL TRIAL: NCT02598713
Title: Validation of Markers for Aspiration for Endotracheal Tube Cuff Leak
Brief Title: Validation of Aspiration Markers in Intubated Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: Aspiration Markers
Record Dates: First submitted 2015-11-02; First posted 2015-11-06 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia; Aspiration
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aspiration Markers (Experimental): Aspiration marker solution will be composed as following: Quinine 83 mg/L suspended in sterile water. After enrollment patients will be challenged with 5 mL of the study solution nebulized in the retropharyngeal space twice a day for two consecutive days.
  Interventions: Drug: Aspiration Marker

INTERVENTIONS:
Drug: Aspiration Marker — Instillation of Quinine suspended in sterile water in the retropharyngeal space of intubated ICU admitted patients for two consecutive days.

SUMMARY:
The goal of this interventional study is to test Quinine as marker of aspiration (endotracheal tube [ETT] cuff leakage) in mechanically ventilated, critically ill patients.

DETAILED DESCRIPTION:
At present there is no standard method for the evaluation of in vivo cuff leak and aspiration. Most of the tested techniques have major pitfalls that render their routine application infeasible. Lacking a practical and reliable marker, any possible intervention aimed at improving cuff seal and ETT performance in order to reduce VAP occurrence is going to be hindered by the inability to truly evaluate its efficacy. Radio-labeled markers are expensive, expose the patient to considerable radiological risk, and require transport to a radiological department, which would expose critically ill patients to additional risk. Dyes have the potential to give useful information about the presence of a cuff leak, but due to persistent staining of secretions, they do not allow continuous monitoring of aspiration. Amylase detection could be a good marker of aspiration, but its ability to detect aspiration is poor even when compared to pepsin. Pepsin and bile acids have the potential to detect some of the aspirations and cuff leaks that happen daily in mechanically ventilated patients, but due to their gastrointestinal nature, they do not offer any kind of information about aspiration of contaminated oropharyngeal secretions. With this research protocol, the investigators would like to validate the use of Quinine suspended in sterile water as marker for determining cuff leakage and aspiration events in an ICU population. Quinine is compound commonly used in food manufacturing. His pharmacokinetic and -dynamic has extensively been studied. The chemical structure of this molecule allows the detection up to pico-molar concentration by spectrophotometry.

The investigators will challenge the oropharyngeal cavity with a known concentration of Quinine suspended in sterile water. The investigators hypothesized that the detection by spectrophotometry of the same substance in the tracheal secretions will prove aspiration.

The investigators specific aims are:

1. To quantify the measurements of Quinine in the tracheal sample and compare with the measurements of Quinine in the oral sample.
2. To assess association between the amount of oropharyngeal aspiration and the development of upper and lower respiratory complications (i.e. ventilator associated pneumonia [VAP], tracheobronchitis, ventilator-associated events, acute respiratory distress syndrome [ARDS], etc.).
3. To determine patient's risk factors associated with oropharyngeal aspiration. The introduction of this new, safe and inexpensive markers for evaluating ETT cuff performance and for detecting aspiration will improve the design of future studies aimed at VAP prevention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to Surgical ICUs (MGH Ellison 4 or Blake 12)
* Patients expected to be intubated for at least 48 hours or longer from the time of enrollment.

Exclusion Criteria:

* High PEEP requirement at enrollment (PEEP higher than 8 cmH2O)
* Diagnosis of ARDS (any severity)
* Status asthmatics
* Current or past participation in another interventional trial conflicting with the present study
* Pregnant women
* Prisoner status
* Patients who had partial or total gastrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Oropharyngeal aspiration: change in concentration of quinine in tracheal samples. | After the beginning of the study, samples will be collected at hours: 0,1 and 24, 25
  The investigators will collect samples of oral and tracheal secretions below the endotracheal tube's cuff. Samples will be centrifuged and the supernatant tested by spectrophotometry. The presence of the study compound in the tracheal samples will be a sign of cuff leak and aspiration. The ratio between the concentration of the study molecules in the oral sample and in the collected samples will be used to give an estimate of leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachussets General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Background] Berra L, Panigada M, De Marchi L, Greco G, Z -Xi Y, Baccarelli A, Pohlmann J, Costello KF, Appleton J, Mahar R, Lewandowski R, Ravitz L, Kolobow T. New approaches for the prevention of airway infection in ventilated patients. Lessons learned from laboratory animal studies at the National Institutes of Health. Minerva Anestesiol. 2003 May;69(5):342-7. PMID 12768164
- [Background] Feldman C, Kassel M, Cantrell J, Kaka S, Morar R, Goolam Mahomed A, Philips JI. The presence and sequence of endotracheal tube colonization in patients undergoing mechanical ventilation. Eur Respir J. 1999 Mar;13(3):546-51. doi: 10.1183/09031936.99.13354699. PMID 10232424
- [Background] Li Bassi G, Luque N, Marti JD, Aguilera Xiol E, Di Pasquale M, Giunta V, Comaru T, Rigol M, Terraneo S, De Rosa F, Rinaudo M, Crisafulli E, Peralta Lepe RC, Agusti C, Lucena C, Ferrer M, Fernandez L, Torres A. Endotracheal tubes for critically ill patients: an in vivo analysis of associated tracheal injury, mucociliary clearance, and sealing efficacy. Chest. 2015 May;147(5):1327-1335. doi: 10.1378/chest.14-1438. PMID 25500677
- [Background] Metheny NA, Clouse RE, Chang YH, Stewart BJ, Oliver DA, Kollef MH. Tracheobronchial aspiration of gastric contents in critically ill tube-fed patients: frequency, outcomes, and risk factors. Crit Care Med. 2006 Apr;34(4):1007-15. doi: 10.1097/01.CCM.0000206106.65220.59. PMID 16484901
- [Background] Mietto C, Pinciroli R, Patel N, Berra L. Ventilator associated pneumonia: evolving definitions and preventive strategies. Respir Care. 2013 Jun;58(6):990-1007. doi: 10.4187/respcare.02380. PMID 23709196